CLINICAL TRIAL: NCT02995239
Title: A Randomized, Open-label, Single Dose, Crossover Study to Compare the Pharmacokinetic Characteristics of CJ-12420 in Healthy Male Volunteers
Brief Title: A Study to Compare the Pharmacokinetic Characteristics of CJ-12420
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_106
Record Dates: First submitted 2016-07-15; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Erosive Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-12420 formulation 1 (Active Comparator): CJ-12420 formulation 1
  Interventions: Drug: CJ-12420 formulation 2
- CJ-12420 formulation 2 (Active Comparator): CJ-12420 formulation 2
  Interventions: Drug: CJ-12420 formulation 1

INTERVENTIONS:
Drug: CJ-12420 formulation 2 — CJ-12420 formulation 2
  Arms: CJ-12420 formulation 1
Drug: CJ-12420 formulation 1 — CJ-12420 formulation 1
  Arms: CJ-12420 formulation 2

SUMMARY:
To compare the pharmacokinetics after administration of different formulation of CJ-12420

DETAILED DESCRIPTION:
The purpose of this study is to compare the pharmacokinetics after a single dose administration of CJ-12420 formulation 1 and formulation 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 19 to 45 years at the screening
* Subject who is over 50kg with BMI between 19 kg/m2 to 28 kg/m2 (inclusive)
* Subject who fully understood after being informed detailed description of clinical trial, written informed consent voluntarily to observe the precautions.

Exclusion Criteria:

* Subject who fall under the criteria below in laboratory test.

  * AST, ALT, ALP, GGT, total bilirubin, BUN, creatinine > UNL x 1.5
* Subject who with low blood pressure with clinical significance at screening test.

  * (systolic blood pressure is less than 90 mmHg or over 140 mmHg, and diastolic blood pressure is less than 50 mmHg or over 90 mmHg)
* Subject who has a medical history of symptomatic GERD, erosive esophagitis or duodenal ulcer, gastric ulcer, barrett's esophagus or zollinger-ellison syndrome.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Assessment of the AUClast | Up to 48 hours

SECONDARY OUTCOMES:
Assessment of the AUCinf | Up to 48 hours
Tmax | Up to 48 hours
t1/2 | Up to 48 hours
Vd/F | Up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, Principal Investigator — Chonbuk university hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided